CLINICAL TRIAL: NCT04844242
Title: A Cross Sectional Study of the Systems Immunology and Viral Diversity of SARS-CoV2 Infection, COVID-19 Disease and Multisystem Inflammatory Syndrome in Children
Brief Title: MISC COVID-19 Study in Pediatric Population
Acronym: COVID-19
Status: Recruiting | Type: Observational
Sponsor: Tuberculosis Research Centre, India (Other Government)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020 034; 2020 034 (Other: NIRT-IEC)
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: SARS-CoV2 Infection; Multisystem Inflammatory Syndrome in Children
MeSH Terms: conditions — COVID-19; pediatric multisystem inflammatory disease, COVID-19 related

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood, nasopharyngeal swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Prior SARS-CoV2 infection as defined by being positive for IgG
- Group 2: COVID-19 disease as defined as children positive by RT-PCR
- Group 3: Children with MIS-C according to the WHO or CDC criteria
- Group 4: Control children who are negative for both RT-PCR and antibody

SUMMARY:
Rationale: Severe Acute Respiratory Syndrome - Coronavirus - 2 (SARS-CoV2) and its related Coronavirus Disease - 19 (COVID-19) has become a health emergency worldwide. The medical community has been concerned since the beginning of the outbreak about the potential impact of COVID-19 in children, especially in those with underlying chronic diseases. Fortunately, COVID-19 has been reported to be less severe in children than in adults. Unfortunately, a new multisystem inflammatory syndrome apparently related to infection with SARS-CoV-2 has recently been reported in older children (known as MIS-C), manifested by severe abdominal pain, cardiac dysfunction and shock. However, the SARS-CoV2 infection and the underlying immunology of COVID-19, its correlation with disease severity and MIS-C in children is not fully explored.

Objectives: To perform systems immunology and strain diversity among SARS-CoV2 and MIS-C infected children.

Study design: Cross sectional study. Study population: Children attending outpatients units and admitted in wards in pediatric hospitals in Chennai.

Main study parameters/endpoints: Immune responses in children with SARS-CoV2 infection and multisystem inflammatory syndrome in children (MIS-C) infection and its association of SARS-CoV2 viral diversity.

DETAILED DESCRIPTION:
Scientific Background:

COVID-19 is a global health crisis. The clinical characteristics, disease progression and outcome in children and young adults appear significantly milder compared to older individuals. Since first being reported in Wuhan, China in December 2019, COVID-19 has rapidly spread, affecting over 200 countries worldwide. Children account for 1-5% of diagnosed COVID-19 cases; although, many infected children may be asymptomatic and therefore not diagnosed without population screening. Most infected children are likely to be secondary cases and acquire the infection after exposure to a COVID-19 positive adult, although there are no longitudinal data to confirm this yet. Intra-family transmission may be important since, an unquantified proportion of children with COVID-19 areasymptomatic and may contribute to transmission. Multiple reports have demonstrated that children and young adults have a milder form of the disease compared to adults. Asymptomatic, mild and moderate infections comprise over 90% of all children who have tested positive for COVID-19 with fewer severe and critical cases (5.9%) compared to adults (18.5%). Given that severe COVID-19 appears very rare in children, an important part of this assessment is ascertaining whether a positive RT-PCR for SARS-CoV-2 is a clinically important factor in explaining the child's condition, or whether more occult pathology may be responsible.

When the COVID-19 pandemic was first reported in Asia and initially spread throughout the globe, pediatricians were grateful that children seemed to be only mildly symptomatic with the infection in most cases. Then, an alarming warning came from the National Health Service in England in April 2020 about cases of older school-aged children and adolescents presenting with fever, hypotension, severe abdominal pain and cardiac dysfunction who tested positive for SARS-CoV-2 infection either by nasopharyngeal RT-PCR assay or by antibody testing. These children had laboratory findings of cytokine storm, including high serum IL-6 levels, and generally required inotropic support to increase cardiac output with rare need for extracorporeal membrane oxygenation. Almost all of these children no longer required intensive care after only a few days and completely recovered, although rare deaths resulted from complications of extracorporeal membrane oxygenation. Case series of children presenting with this condition have now been reported from the UK, Italy, Spain, France and Switzerland, and the United States. The Centers for Disease Control and Prevention (CDC) has developed a case definition for use in the United States and has termed the condition multisystem inflammatory syndrome in children (MIS-C). If MIS-C is indeed related to infection with SARS-CoV-2, the pathophysiological mechanism of disease is unclear.

Very few studies have addressed the immune responses to SARS-CoV2 (either humoral or cell mediated immunity) in children. It is therefore necessary to study the immune responses in asymptomatic infections, prior infections and MIS-C to understand the pathogenesis of the disease.

Whole-genome sequencing of pathogens, especially viruses, is a powerful tool to generate rapid information on outbreaks, resulting in effective understanding of the introduction of the infection, dynamics of transmission, and impact of informed outbreak control decisions. In- deed, genomic data can be used to identify pathogen genes interacting with the host and allows characterisation of the more evolutionary constrained regions of a pathogen genome, which should be preferentially targeted to avoid rapid drug and vaccine escape mutants. (1). As the SARS-CoV-2 virus races around the world across the different population, there needs to be a consolidated effort to understand the divergence of demographically distributed strains. Since the transmission of SARS-CoV-2 is subject to the extent of human interaction, the insights from the correlation of genetic diversity would give vital information to tackle this transmission.

Recent published studies have reported that when comparing the 305 Indian SARS-CoV-2 genomes, a number of nucleotide variants or segregating sites being identified. Recent literature report that there is the presence of multiple lineages of SARS-CoV-2 in India in different geographic regions. 20A and 20B together (belonging to the former haplotype of A2a) are the predominant haplotypes at pan India level and in each region. Interestingly, the haplotypes were differentially distributed in different regions. While the 20A were most abundant in Northern and Eastern India, 20B was found to be the most abundant haplotype in Western and Southern India. The ancestral haplotypes of 19A and 19B were mostly found in Northern and Eastern India, with 19B being the most abundant in the latter region. While multiple haplotypes were introduced during the early part of the outbreak in March-May 2020, the 20A, B and C haplotypes (A2a) became the predominant haplotypes in all regions by June 2020. However, there are no studies that have characterised the viral diversity in this pediatric population and its association with immunological response and disease severity, in SARS-CoV-2 infected children.

Study objectives:

* To perform systems immunology of SARS-CoV2 infection, COVID-19 disease and MIS-C in children
* To identify the SARS-CoV2 viral diversity in the pediatric population and correlate with immune responses and disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 to 15 years of age
* Willing to provide informed consent (parents)/assent
* For Group 1 - Positive or Negative for COVID-19 by RT-PCR but positive for SARS-CoV2 IgG
* For Group 2 - Positive for COVID-19 by RT-PCR but negative for SARS-CoV2 IgG
* For Group 3 - Positive for COVID-19 by RT-PCR or positive for SARS-CoV2 IgG antibody
* For Group 4 - Control children who are negative for both RT-PCR and IgG antibody

Exclusion Criteria:

* Severely immunocompromised or anemic (WHO criteria in children) or malnourished
* History of any illness or condition which, in the investigator's judgment, may substantially increase the risk associated with the participant's participation in the protocol, or compromise the scientific objectives

Ages: 1 Year to 15 Years | Sex: All
Age Groups: Child
Study Population: Children attending outpatient clinics and admitted in the wards of Institute Of Child Health and Hospital for Children, Rainbow Childrens Hospital and Dr. Mehta's Childrens Hospitals, Chennai.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterization of immune responses | 6 months
  Immune responses in children with SARS-CoV2 infection and multisystem inflammatory syndrome in children (MIS-C) infection and its association of SARS-CoV2 viral diversity

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute for Research in Tuberculosis, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rajamanickam A, Nathella PK, Venkataraman A, Varadarjan P, Kannan S, Pandiarajan AN, Renji RM, Elavarasan E, Thimmaiah A, Sasidaran K, Krishnamoorthy N, Natarajan S, Ramaswamy G, Sundaram B, Putlibai S, Hissar S, Selladurai E, Uma Devi KR, Nutman TB, Babu S. Unique cellular immune signatures of multisystem inflammatory syndrome in children. PLoS Pathog. 2022 Nov 2;18(11):e1010915. doi: 10.1371/journal.ppat.1010915. eCollection 2022 Nov. PMID 36322537